CLINICAL TRIAL: NCT05195216
Title: Psychosocial Factors and Quality of Life in the Effect of Fear of COVID-19 With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Elif Kabasakal (Other)
Responsible Party: Sponsor-Investigator, Elif Kabasakal, ekabasakal, Medipol University
Organization: Medipol University (Other)
Other Study IDs: MedipolU-KABASAKAL-001
Record Dates: First submitted 2022-01-13; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- individuals with cystic fibrosis
  Interventions: Behavioral: Survey Form, The Hospital Anxiety and Depression Scale, The Fear of COVID-19 Scale,World Health Organization Quality of Life Scale- Bref Form
- healthy individuals
  Interventions: Behavioral: Survey Form, The Hospital Anxiety and Depression Scale, The Fear of COVID-19 Scale,World Health Organization Quality of Life Scale- Bref Form

INTERVENTIONS:
Behavioral: Survey Form, The Hospital Anxiety and Depression Scale, The Fear of COVID-19 Scale,World Health Organization Quality of Life Scale- Bref Form — Online questionnaires were administered to individuals.

SUMMARY:
The purpose of this study; The COVID-19 pandemic is to investigate the effects of COVID-19 fear levels of patients with cystic fibrosis on the psychosocial and quality of life levels of individuals.

DETAILED DESCRIPTION:
After individuals were informed about the study, it was administered to individuals who gave written informed consent.This study was carried out on individuals with cystic fibrosis and healthy individuals who meet the eligibility requirements, through online forms.

ELIGIBILITY:
Inclusion Criteria:

* be 16 years of age or older
* Having been diagnosed with Cystic Fibrosis
* Volunteering to participate in the research

Exclusion Criteria:

* Being mentally incapable of successfully applying the scales to be applied for evaluation purposes
* Being treated with sedative and antiepileptic drugs
* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 64 individuals with cystic fibrosis and 70 healthy individuals participated in the study.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
fear of covid-19 | November- December/2021
  COVID-19 Fear Scale: This scale is a one-dimensional instrument consisting of seven items with robust psychometric properties that measure fear of COVID-19. It has a 5-point Likert-type rating system (1: Strongly disagree, 5: Strongly agree). It is reliable and valid in assessing fear of COVID-19 among the general population. Turkish validity and reliability of the scale were ensured.

SECONDARY OUTCOMES:
psychosocial factors | November-December/2021November-December/2021
  Hospital Anxiety and Depression Scale (HADS): The scale consists of 14 items. 7 of these items measure anxiety and 7 of them measure depression symptoms. The items in the scale are evaluated with a 4-point Likert scale and are based on a scoring system between 0-3.

OTHER OUTCOMES:
quality of life assessment | November-December/2021November-December/2021
  It is an internationally comparable assessment tool developed by the World Health Organization. The scale evaluates the level of quality of life. The scale consists of 26 items. The Turkish version of WHOQOL-Bref consists of 27 items. Question 27 has been added to the Turkish version of the scale as a national environmental field and is used only in national studies. The scale includes the areas of physical health, psychological health, social relations, environment and national environment. It has a 5-point likert-type rating system. The score of each area is important on its own. Higher scores in each area indicate better quality of life. The first two questions of the quality of life scale are not included in the scoring and are evaluated separately. The number of questions, which was 26 in the original of the scale, is used as 27 in the Turkish version.

CONTACTS AND LOCATIONS:
Locations (1):
- Elif Kabasakal, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No